CLINICAL TRIAL: NCT00413257
Title: Study of the Effects of Nefopam on Hyperalgesia Following Sternotomy in Cardiac Surgery
Brief Title: Effects of Nefopam on Hyperalgesia After Cardiac Surgery
Acronym: NefalCard
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7813; 2005-033
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Hyperalgesia; Pain, Postoperative; Pain, Chronic Disease
Keywords: Postoperative Hyperalgesia; cardiac Surgical Procedures; Nefopam; Randomized Controlled Trials; Pain and chronic disease
MeSH Terms: conditions — Hyperalgesia; Pain, Postoperative; Pain; Chronic Disease | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): nefopam infusion will start before the surgical incision, at the induction time of anesthesia and will be continued until postoperative H48
  Interventions: Drug: Nefopam
- 2 (Experimental): nefopam administration will start at the end of the surgery and will be continued until postoperative H48
  Interventions: Drug: néfopam
- 3 (Placebo Comparator): control group that will receive a placebo from the induction time of anesthesia until H48
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Nefopam — 0,3mg/kg IV bolus preoperative and 65 µg/kg/h during H48 postoperative
  Arms: 1
Drug: néfopam — bolus Néfopam (0,3mg/kg) during 10 min at the end of surgery and 65 µg/kg/h during postoperative H48
  Arms: 2
Drug: Placebo comparator — bolus NaCl during 10 min at the end of surgery and during postoperative H48
  Arms: 3

SUMMARY:
Postoperative pain after major surgery is consecutive not only to the nociceptive inputs coming from the surgical lesion, but also to peripheral and central neuronal sensitization. This lead to postoperative hyperalgesia and allodynia that are enhanced by the per operative use of high opioid doses. Anti-NMDA drugs have been reported as able to reduce this sensitization process and then to decrease acute morphine tolerance during the postoperative period. Nefopam has been lately shown to combine in experimental trials analgesic and anti hyperalgesic effects. The aim of this study is to compare anti-hyperalgesic effects of nefopam given either before incision and continuously for the following 48hours or starting from the end of the surgery and given for 48hours to a control group that would receive placebo for 48hours. Postoperative analgesia will be based on morphine PCA. Pain scores, hyperalgesia, allodynia, postoperative morphine consumption, and development of chronic pain will be the main criteria that will be evaluated during this study

DETAILED DESCRIPTION:
Introduction :

Postoperative pain is not only a consequence of the surgical lesion, but is also related to sensitization processes that appear in peripheral and central nerves. This sensitization induce clinically hyperalgesia and allodynia. From an experimental viewpoint it comes mainly from a central activation of NMDA receptors in neurons that conduct the nociceptive message.

Recent studies have shown that high-dose opioids were able, via NMDA receptors, to enhance postoperative hyperalgesia and to increase pain scores and morphine consumption after surgery. Nevertheless per operative use of opioid is still necessary to avoid per operative stress and systemic consequence of the surgical stimulation.

Some drugs (ketamine, nitrous oxide…) succeeded in reducing postoperative hyperalgesia and pains scores and acute morphine tolerance. They also were able to decrease pain chronicization.

Nefopam, well known as an analgesic since the 80's, presents both analgesic and anti hyperalgesic properties as lately demonstrated in experimental trials. Nevertheless these anti hyperalgesic properties have never been evaluated in humans scheduled for cardiac surgery. Nefopam administration could reduce acute morphine tolerance and could enhance postoperative pain management by reducing sensitization processes and hyperalgesia.

Objective :

The main purpose of this clinical trial will be to evaluate in patients scheduled for cardiac surgery with sternotomy the nefopam effects on the nociceptive threshold evaluated with dynamic Von Frey mechanical stimulation.

The secondary objectives will evaluate static hyperalgesia, postoperative pain scores, morphine consumption, cognitive functions, and development of chronic pain and dysesthesia.

Methods :

Prospective, randomized, double-blind study that will compare three parallel groups that will receive the same per operative anesthesia except for the nefopam doses.

Group 1: nefopam infusion will start before the surgical incision, at the induction time of anesthesia and will be continued until postoperative H48. Group 2: nefopam administration will start at the end of the surgery and will be continued until postoperative H48. Group 3: control group that will receive a placebo from the induction time of anesthesia until H48. All patients will receive postoperatively morphine infusion following the Patient Controlled Analgesia concept.

Number of patients to be included : 90 Duration of the study : 2 years Start : second semester of 2006

Expected result :

Reduction of the extend of hyperalgesia around the wound evaluated with dynamic Von Frey mechanical stimulation more than 20%.

ELIGIBILITY:
Inclusion Criteria:

* 55-75 years old
* ASA score: 1-3
* Patients scheduled for Cardiac surgery with median sternotomy for : single valve replacement or Bentall or Benson or Tyron David surgery, single or multiple Cardiac Artery Bypass Grafting (CABG) , combined surgery (valve replacement + CABG) without preoperative risk of postoperative complications
* Informed consent obtained from the patient

Exclusion Criteria:

* Drug or alcohol abuse history
* Analgesic or opioid consumption within the 12hs preceding the surgery
* Chronic use of analgesic drugs or history of chronic pain
* Convulsion or epilepsy history
* Glaucoma history
* Disability to understand morphine PCA use
* Allergy to nefopam

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Nociceptive threshold evaluated with Von Frey mechanical dynamic stimulation. This will start 10cm far from the wound on a perpendicular line to the wound and will be conducted by 1cm step to the wound until the patient explains the stimulation | H 24

SECONDARY OUTCOMES:
static hyperalgesia with Von Frey stimulation 1cm far from the middle of the wound, on the right side of the wound. | 1, 2, 4 and 7 days after intervention
Morphine consumption | over the 48 H postoperative
Pain scores evaluation | Acute pain (1, 2, 4 and 7 days after intervention) / Chronic Pain (3, 6 and 12 month)
Cognitive functions evaluation | 1, 2, 4 and 7 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RICHEBE, Dr, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Département d'Anesthésie-Réanimation II - Hôpital cardiologique - Groupe Hospitalier Sud, CHU de Bordeaux - 4, Av de Magellan, Pessac, France

REFERENCES:
- [Derived] Richebe P, Picard W, Rivat C, Jelacic S, Branchard O, Leproust S, Cahana A, Janvier G. Effects of nefopam on early postoperative hyperalgesia after cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Jun;27(3):427-35. doi: 10.1053/j.jvca.2012.08.015. Epub 2012 Oct 12. PMID 23063945